CLINICAL TRIAL: NCT02065336
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Determine the Depth and Duration of Hepatitis B Surface Antigen (HBsAg) Reduction After a Single Intravenous Dose of ARC-520 in Combination With Entecavir in Patients With Chronic Hepatitis B Virus (HBV) Infection, Followed by a Two-dose Open-label Cohort and Three Open-label Single-dose Cohorts in Treatment Naïve Patients, Including a Multi-dose Open-label Extension at a Single Center
Brief Title: A Multicenter Study to Determine the Depth and Duration of Hepatitis B Surface Antigen (HBsAg) Reduction After Single or Multiple Doses of ARC-520, in Combination With Entecavir in Patients With Chronic Hepatitis B Virus (HBV) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Heparc-2001
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B, Chronic
Keywords: HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis | interventions — ARC-520; entecavir; Chlorpheniramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- ARC-520 Cohort 1 (Experimental): a single intravenous (IV) dose of double-blind ARC-520 Injection 1.0 mg/kg in combination with entecavir administered to participants with HBeAg-negative immune active chronic HBV infection
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 2 (Placebo Comparator): a single IV dose of double-blind ARC-520 Injection 2.0 mg/kg in combination with entecavir administered to participants with HBeAg-negative immune active chronic HBV infection
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 3 (Experimental): a single IV dose of double-blind ARC-520 Injection 3.0 mg/kg in combination with entecavir administered to participants with HBeAg-negative immune active chronic HBV infection
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 4 (Experimental): a single IV dose of double-blind ARC-520 Injection 4.0 mg/kg in combination with entecavir administered to participants with HBeAg-negative immune active chronic HBV infection
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 5 (Experimental): a single IV dose of double-blind ARC-520 Injection 4.0 mg/kg in combination with entecavir administered to participants with HBeAg-positive immune active chronic HBV infection
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- Placebo Normal Saline Cohorts 1-5 (Experimental): a single IV dose of double-blind normal saline in combination with entecavir administered to participants with HBeAg-negative or -positive immune active chronic HBV infection
  Interventions: Drug: Placebo; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 6 (Experimental): two IV doses of open-label ARC-520 2.0 mg/kg administered to participants with HBeAg-positive immune active chronic HBV
  Interventions: Drug: ARC-520; Drug: chlorpheniramine
- ARC-520 Cohort 7 (Experimental): a single IV dose of open-label ARC-520 4.0 mg/kg administered to treatment-naïve, HBeAg-negative or -positive participants with chronic hepatitis B (CHB)
  Interventions: Drug: ARC-520; Drug: chlorpheniramine
- ARC-520 Cohort 8 (Experimental): open-label multi-dose extension cohort: multiple IV doses of open-label ARC-520 (4.0 mg/kg every [Q]4 weeks) administered to HBeAg-negative participants with CHB receiving chronic entecavir therapy who completed Cohorts 1 through 4
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 9 (Experimental): open-label multi-dose extension cohort: multiple IV doses of open-label ARC-520 (4.0 mg/kg Q6 weeks or Q8 weeks) administered to HBeAg-positive participants with CHB receiving chronic entecavir therapy who completed Cohorts 5 or 6
  Interventions: Drug: ARC-520; Drug: entecavir; Drug: chlorpheniramine
- ARC-520 Cohort 10 (Experimental): open-label multi-dose extension cohort: multiple IV doses of open-label ARC-520 (4.0 mg/kg Q4 weeks) administered to a mixed cohort (HBeAg-negative and -positive participants) who were naïve (within the last 6 months) to entecavir treatment and completed Cohort 7
  Interventions: Drug: ARC-520; Drug: chlorpheniramine
- ARC-520 Cohort 11 (Experimental): a single IV dose of open-label ARC-520 5.0 mg/kg administered to treatment-naïve, HBeAg-positive participants with CHB
  Interventions: Drug: ARC-520; Drug: chlorpheniramine
- ARC-520 Cohort 12 (Experimental): a single IV dose of open-label ARC-520 6.0 mg/kg administered to treatment-naïve, HBeAg-positive participants with CHB
  Interventions: Drug: ARC-520; Drug: chlorpheniramine

INTERVENTIONS:
Drug: ARC-520
  Arms: ARC-520 Cohort 1; ARC-520 Cohort 10; ARC-520 Cohort 11; ARC-520 Cohort 12; ARC-520 Cohort 2; ARC-520 Cohort 3; ARC-520 Cohort 4; ARC-520 Cohort 5; ARC-520 Cohort 6; ARC-520 Cohort 7; ARC-520 Cohort 8; ARC-520 Cohort 9
Drug: Placebo
  Arms: Placebo Normal Saline Cohorts 1-5
Drug: entecavir
  Other Names: Baraclude
  Arms: ARC-520 Cohort 1; ARC-520 Cohort 2; ARC-520 Cohort 3; ARC-520 Cohort 4; ARC-520 Cohort 5; ARC-520 Cohort 8; ARC-520 Cohort 9; Placebo Normal Saline Cohorts 1-5
Drug: chlorpheniramine — In all cohorts, each participant received an 8 mg dose of oral chlorpheniramine 2 hours prior to each administration of ARC-520 Injection.

SUMMARY:
The purpose of this study is to determine whether ARC-520 in combination with entecavir is effective in the treatment of patients with chronic HBV Infection.

DETAILED DESCRIPTION:
Treatment with ARC-520 for injection is expected to reduce all HBV proteins and replicative intermediates via ribonucleic acid (RNA) interference. The magnitude of the reduction and duration of effect will depend on the dose. Since to date ARC-520 has not been administered to patients with chronic HBV infection, the effective therapeutic dose in patients with chronic HBV infection is unknown. This study is designed to assess the antiviral activity of ARC-520, especially its effect on HBsAg, in patients with chronic HBV infection at different dose levels.

This is a multicenter, randomized, double-blind, placebo-controlled, single-dose escalation study of ARC 520 in combination with entecavir administered to participants with hepatitis B virus e antigen (HBeAg)-negative (Cohorts 1 through 4) or HBeAg-positive (Cohort 5) immune active, chronic HBV infection, followed by a two-dose open-label cohort (Cohort 6), three open-label single-dose cohorts in treatment-naïve participants (Cohorts 7, 11 and 12) and an open-label multi-dose extension study (Cohorts 8, 9, 10). Cohort 6 will investigate ARC-520 in combination with entecavir administered in two doses to participants with HBeAg-positive immune-active chronic HBV infection. Cohorts 7, 11 and 12 will enroll treatment-naïve participants. Cohort 8 will only enroll participants previously completing Cohorts 1-4. Cohort 9 will only enroll participants previously completing Cohort 5 or 6. Cohort 10 will only enroll participants previously completing Cohort 7.

Participants will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate, and temperature), weight, adverse events (AEs), 12-lead electrocardiograms (ECGs), concomitant medication, blood sample collection for hematology, coagulation, chemistry, pharmacokinetic (PK) and exploratory pharmacodynamic (PD) measures, urinalysis, HBV serology, HBV genotyping and sequencing, follicle stimulating hormone (FSH) testing and pregnancy testing for females of childbearing potential. Clinically significant changes including AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the participant is lost to follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of HBeAg negative and immune active chronic HBV infection (Cohorts 1-4, 8)
* Diagnosis of HBeAg positive and immune active chronic HBV infection (Cohorts 5-6, 9)
* Diagnosis of HBeAg negative or HBeAg positive and immune active or tolerant chronic HBV infection (Cohorts 7, 10, 11 & 12)
* Patients with > 6 months of continuous, 0.5 mg/day oral entecavir, and a willingness to continue taking entecavir throughout the study (Cohorts 1-6, 8-9).
* Patients naive to entecavir (never on entecavir or on entecavir <30 days prior to screening) and a willingness to take entecavir and willingness to continue taking entecavir throughout the study (Cohorts 7, 11 & 12).

Key Exclusion Criteria:

* Female patients that have a positive pregnancy test or are lactating.
* Acute signs of hepatitis/other infection (eg, moderate fever, jaundice, nausea, vomiting, and abdominal pain) evident within 4 weeks of screening and/or at the screening examination.
* Patients with antiviral therapy other than entecavir within 3 months of screening or prior treatment with interferon or a toll receptor agonist in the last 5 years.
* Use within the last 6 months or an anticipated requirement for anticoagulants, corticosteroids, immunomodulators, or immunosuppressants.
* Has any history of autoimmune disease especially autoimmune hepatitis.
* Has human immunodeficiency virus (HIV) infection, as shown by the presence of anti-HIV antibody (sero-positive).
* Is sero-positive for hepatitis C virus (HCV), and/or a history of delta virus hepatitis.
* Has a history of allergy to bee venom or history of hypersensitivity reaction requiring an emergency visit to a physician or hospital and/or requirement for treatment with steroids and/or epinephrine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Given, MD, Study Chair — Arrowhead Pharmaceuticals, Inc.
Locations (2):
- Hong Kong (2):
  - Research Site 1, Pokfulam
  - Research Site 2, Shatin

REFERENCES:
- [Derived] Yuen MF, Wong DK, Schluep T, Lai CL, Ferrari C, Locarnini S, Lo RC, Gish RG, Hamilton J, Wooddell CI, Mak LY, Given BD. Long-term serological, virological and histological responses to RNA inhibition by ARC-520 in Chinese chronic hepatitis B patients on entecavir treatment. Gut. 2022 Apr;71(4):789-797. doi: 10.1136/gutjnl-2020-323445. Epub 2021 Mar 12. PMID 33712437

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were enrolled in Cohorts 8, 11, or 12. Cohort 9 (n=2) and Cohort 10 (n=8) enrolled participants who previously completed treatment in other cohorts.
Period: Main Study
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | Placebo Normal Saline Cohorts 1-5 | ARC-520 Cohort 9 | ARC-520 Cohort 10
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | Placebo Normal Saline Cohorts 1-5 | ARC-520 Cohort 9 | ARC-520 Cohort 10
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- ARC-520 Cohort 1: a single IV dose of double-blind ARC-520 Injection 1.0 mg/kg in combination with entecavir administered to participants with HBeAg-negative immune active chronic HBV infection
- Total: Total of all reporting groups
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | Placebo Normal Saline Cohorts 1-5 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (8.22) | 43.0 (4.15) | 42.0 (1.79) | 39.8 (2.04) | 39.5 (7.23) | 33.3 (4.23) | 39.8 (10.12) | 44.4 (9.09) | 41.4 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 1 | 2 | 3 | 5 | 2 | 20
  Male | 4 | 4 | 3 | 5 | 4 | 3 | 7 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Over Time in Quantitative Hepatitis B Surface Antigen (HBsAG)
Time Frame: Baseline, through Day 85 (Cohorts 1-7) and through 24 weeks post-last dose (last dose: Day 85 Cohort 9; Day 253 Cohort 10)
Population: Pharmacodynamic (PD) Population: all participants who received at least 1 dose of study drug and had evaluable data from at least one postdose PD assessment according to the treatment the participants were assigned.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | Placebo Normal Saline Cohorts 1-5 | ARC-520 Cohort 9 | ARC-520 Cohort 10
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 8
IU/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Day 1 |  |  |  |  |  |  |  |  |  | -19222 (27217)
  Day 3: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 0
  Day 3 | -554.8 (861.86) | -1194.0 (2083.72) | -1003.6 (949.36) | -1501.0 (1930.12) | -1664.7 (2375.62) | -948.0 (1016.31) | -12401.1 (17661.02) | 43.3 (267.60) |  |
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 0
  Day 8 | -928.1 (1285.26) | -2179.2 (3170.68) | -884.3 (1296.49) | -2591.2 (3304.72) | -1789.8 (2101.23) | -1344.0 (1319.66) | -20123.8 (29795.99) | 42.2 (568.32) |  |
  Day 15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0 | 12 | 10 | 0 | 0
  Day 15 | -1055.1 (1900.89) | -2260.8 (4022.82) | -470.8 (2025.31) | -3069.0 (3923.45) | -1672.8 (1892.73) |  | -22915.6 (34381.59) | 236.6 (321.17) |  |
  Day 22: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 0
  Day 22 | -1225.4 (1967.15) | -2266.2 (3868.90) | -204.3 (2077.12) | -2978.8 (3536.73) | -1951.7 (2819.85) | -1553.7 (1596.05) | -23872.7 (35753.39) | 115.1 (594.38) |  |
  Day 29 | -579.1 (352.71) | -1826.3 (2618.78) | 93.3 (2425.68) | -2972.8 (3506.01) | -1964.3 (2501.62) | -1532.3 (1500.40) | -24148.3 (36256.02) | 168.8 (460.59) |  | -22617 (32653)
  Day 43: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 0
  Day 43 | -1020.1 (1252.98) | -1288.8 (1498.60) | -1471.8 (1625.30) | -3219.8 (3601.70) | -1939.7 (2277.79) | -1566.8 (1290.46) | -23932.0 (35929.80) | 58.3 (411.60) |  |
  Day 57: number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 12 | 10 | 0 | 8
  Day 57 |  | -1056.7 (773.69) | -2330.1 (1676.50) | -2813.0 (2665.97) | -1536.0 (1373.46) | -1370.7 (872.64) | -22658.4 (34292.84) | 156.1 (527.40) |  | -22840 (32239)
  Day 85 | -670.1 (1825.99) | -542.8 (1815.34) | -2119.3 (1717.17) | -926.3 (1406.29) | -537.5 (1901.16) | -791.0 (457.04) | -20827.2 (31753.76) | 225.4 (393.81) |  | -23305 (32455)
  Day 113: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Day 113 |  |  |  |  |  |  |  |  |  | -23205 (32362)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Day 141 |  |  |  |  |  |  |  |  |  | -23182 (32379)
  Day 169: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Day 169 |  |  |  |  |  |  |  |  |  | -26481 (33649)
  Day 197: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Day 197 |  |  |  |  |  |  |  |  |  | -30234 (34097)
  Day 225: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Day 225 |  |  |  |  |  |  |  |  |  | -1249 (1273)
  Day 253: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Day 253 |  |  |  |  |  |  |  |  |  | -643 (905)

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. An SAE is any AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction.Events were categorized as mild, moderate or severe. TEAEs were defined as all AEs starting or worsening after commencement of treatment with investigational product. A treatment-related TEAE was one whose relationship to treatment was noted as unlikely, possibly, or probably related.
Time Frame: through Day 85 (Cohorts 1-7) and through 24 weeks post-last dose (last dose: Day 85 Cohort 9; Day 225 Cohort 10)
Population: Safety Population: all participants who received any amount of study drug or placebo, and had at least 1 postdose safety assessment. Data for Cohort 9 was not analyzed or summarized due to limited enrollment.
Measure: Count of Participants; unit: Participants
Groups:
- ARC-520 Cohort 7: a single IV dose of open-label ARC-520 4.0 mg/kg administered to treatment-naïve, HBeAg-negative or -positive participants with CHB
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 9 | ARC-520 Cohort 10 | Placebo Normal Saline Cohorts 1-5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 2 | 8 | 10
Participants
  Any TEAE | 1 | 4 | 1 | 0 | 1 | 1 | 1 | 1 | 7 | 0
  Any mild TEAE | 1 | 3 | 1 | 0 | 1 | 1 | 1 | 1 | 7 | 0
  Any moderate TEAE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any severe TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
  Any TEAE leading to discontinuation of treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any life-threatening SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Negative Bee Venom Allergy Test Results at Baseline, Day 29, and Day 85
Description: Bee venom allergy tests were used to assess immunoglobulin E (IgE) in Cohorts 1-7. Analysis values less than 0.35 kU/L were taken as negative.
Time Frame: Baseline, Day 29, Day 85
Population: Safety Population: all participants who received any amount of study drug or placebo, and had at least 1 postdose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- ARC-520 Cohort 6: two IV doses of open-label ARC-520 2.0 mg/kg administered to participants with HBeAg-positive immune-active chronic HBV
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | Placebo Normal Saline Cohorts 1-5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10
Participants
  Baseline | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10
  Day 29 | 6 | 6 | 6 | 6 | 6 | 6 | 11 | 10
  Day 85 | 6 | 6 | 6 | 6 | 6 | 6 | 11 | 10

4. Secondary Outcome: Change From Baseline in Entecavir Plasma Trough Concentration, Cohorts 1-7
Time Frame: Baseline, Days 1, 2, 3, 8, 15, 22, 29
Population: Pharmacokinetic (PK) Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ARC-520 Cohorts 4 and 5: a single IV dose of double-blind ARC-520 Injection 4.0 mg/kg in combination with entecavir administered to participants with HBeAg-negative immune active chronic HBV infection or participants with HBeAg-positive immune active chronic HBV infection
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohorts 4 and 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | Placebo Normal Saline Cohorts 1-5
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 6 | 12 | 10
ng/mL
  Day 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 2 | 0.06 (0.05) | 0.06 (0.08) | 0.13 (0.08) | 0.12 (0.10) | -0.91 (1.59) | 0.16 (0.04) | -0.31 (0.89)
  Day 3 | -0.02 (0.02) | -0.06 (0.09) | -0.06 (0.06) | 0.12 (0.63) | -1.04 (1.58) | 0.15 (0.03) | -0.29 (0.88)
  Day 8 | -0.01 (0.07) | -0.09 (0.08) | -0.09 (0.13) | -0.03 (0.18) | -1.01 (1.60) | 0.45 (0.76) | -0.30 (0.90)
  Day 15 | 0.01 (0.05) | -0.03 (0.12) | -0.03 (0.06) | 0.00 (0.18) | -1.01 (1.63) | 0.32 (0.11) | -0.10 (1.14)
  Day 22 | 0.04 (0.06) | -0.02 (0.14) | -0.03 (0.09) | 0.00 (0.13) | -1.00 (1.58) | 0.33 (0.11) | -0.30 (0.89)
  Day 29 | 0.00 (0.06) | -0.01 (0.11) | 0.01 (0.07) | 0.00 (0.15) | -1.00 (1.61) | 0.36 (0.11) | -0.30 (0.89)

5. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
µg*hr/mL
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 79.1 (8.28) | 185 (61.2) | 212 (34.7) | 318 (82.3) | 349 (45.2)
  AD0010 | 93.0 (9.11) | 190 (43.2) | 301 (43.9) | 370 (80.5) | 412 (47.5)

6. Secondary Outcome: Pharmacokinetics of ARC-520 of ARC-520 Product Constituents AD0009 and AD0010: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Quantifiable Plasma Concentration (AUClast), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
µg*hr/mL
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 81.4 (9.25) | 196 (66.3) | 218 (37.1) | 326 (87.3) | 356 (47.4)
  AD0010 | 97.6 (9.77) | 205 (50.2) | 317 (50.7) | 385 (88.0) | 434 (53.3)

7. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf), Cohorts 1-5 Only
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
µg*hr/mL
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 81.4 (9.26) | 196 (66.3) | 218 (37.2) | 326 (87.4) | 356 (47.4)
  AD0010 | 97.8 (9.80) | 207 (51.1) | 318 (51.2) | 386 (88.6) | 435 (53.8)

8. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Maximum Observed Plasma Concentration (Cmax), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
µg/mL
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 13.7 (2.42) | 26.4 (6.84) | 33.5 (1.78) | 54.8 (9.59) | 58.2 (5.88)
  AD0010 | 12.7 (2.07) | 22.5 (2.74) | 39.7 (2.60) | 50.5 (10.6) | 52.4 (6.44)

9. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Clearance (CL), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mL/hr/kg
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 6.21 (0.724) | 5.58 (1.84) | 7.11 (1.56) | 6.47 (1.51) | 5.70 (0.781)
  AD0010 | 5.16 (0.522) | 5.08 (1.19) | 4.84 (0.952) | 5.41 (1.19) | 4.65 (0.586)

10. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Apparent Volume of Distribution During the Terminal Phase (Vz), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mL/kg
  AD0009 | 39.5 (4.13) | 43.2 (15.8) | 45.7 (5.72) | 39.0 (7.27) | 35.4 (4.06)
  AD0010 | 39.4 (5.01) | 46.1 (9.99) | 37.1 (2.52) | 37.9 (5.83) | 36.9 (3.18)

11. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Volume in Steady State (Vss), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mL/kg
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 39.6 (6.05) | 45.8 (11.6) | 45.3 (3.60) | 39.6 (6.31) | 35.3 (3.57)
  AD0010 | 40.7 (6.01) | 46.7 (8.22) | 38.1 (2.08) | 39.8 (6.36) | 38.5 (4.21)

12. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Terminal Elimination Rate Constant (Kel), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
1/hr
  AD0009 | 0.157 (0.0115) | 0.132 (0.0242) | 0.154 (0.0135) | 0.165 (0.0120) | 0.161 (0.00614)
  AD0010 | 0.132 (0.0131) | 0.111 (0.0188) | 0.130 (0.0180) | 0.142 (0.0164) | 0.126 (0.00793)

13. Secondary Outcome: Pharmacokinetics of ARC-520 Product Constituents AD0009 and AD0010: Terminal Elimination Half-Life (t1/2), Cohorts 1-5
Time Frame: Day 1 predose, immediately prior to the end of infusion, 0.5, 1, 3, 6, 24, and 48 hours postdose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours
  AD0009: number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
  AD0009 | 4.38 [4.06 to 4.96] | 5.36 [4.16 to 7.00] | 4.64 [3.87 to 4.90] | 4.18 [3.92 to 4.87] | 4.32 [4.14 to 4.60]
  AD0010 | 5.29 [4.76 to 6.19] | 6.32 [5.09 to 7.94] | 5.48 [4.26 to 6.41] | 4.79 [4.32 to 6.15] | 5.36 [5.16 to 6.02]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Day 85 (Cohorts 1-7) and through 24 weeks post-last dose (last dose: Day 85 Cohort 9; Day 225 Cohort 10)
Arm/Group | ARC-520 Cohort 1 | ARC-520 Cohort 2 | ARC-520 Cohort 3 | ARC-520 Cohort 4 | ARC-520 Cohort 5 | ARC-520 Cohort 6 | ARC-520 Cohort 7 | ARC-520 Cohort 9 | ARC-520 Cohort 10 | Placebo Normal Saline Cohorts 1-5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/2 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 4/6 | 1/6 | 0/6 | 1/6 | 1/6 | 1/12 | 1/2 | 7/8 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARC-520 Cohort 1 (N=6) | ARC-520 Cohort 2 (N=6) | ARC-520 Cohort 3 (N=6) | ARC-520 Cohort 4 (N=6) | ARC-520 Cohort 5 (N=6) | ARC-520 Cohort 6 (N=6) | ARC-520 Cohort 7 (N=12) | ARC-520 Cohort 9 (N=2) | ARC-520 Cohort 10 (N=8) | Placebo Normal Saline Cohorts 1-5 (N=10)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The ARC-520 Injection development program was terminated early for regulatory and business reasons secondary to findings occurring in a non-clinical toxicology study. Program termination was not due to safety findings in humans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No